CLINICAL TRIAL: NCT03224208
Title: VECODUE A Phase II Trial of Vemurafenib Plus Cobimetinib in Patients Treated With Prior First-line Systemic Immunotherapy for Inoperable Locally Advanced or Metastatic Melanoma
Brief Title: Vemurafenib Plus Cobimetinib in Advanced or Metastatic Melanoma Patients
Acronym: VECODUE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrolment rate
Sponsor: Fondazione Melanoma Onlus (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VECODUE
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Melanoma; Melanoma (Skin); Melanoma Stage
Keywords: melanoma; advanced; vemurafenib; cobimetinib
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Vemurafenib will be orally adminitered at 960 mg b.i.d. on Days 1-28. Cobimetinib will be given orally at 60 mg qd on Days 1-21 of each 28-day treatment cycle until disease progression.
  Treatments will be continued until the development of progressive disease (as per Investigator assessment), unacceptable toxicity, consent withdrawal, death, reasons deemed by the treating physician or study termination by the Sponsor.
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib

INTERVENTIONS:
Drug: Vemurafenib — Vemurafenib will be orally adminitered at 960 mg b.i.d. on Days 1-28
Drug: Cobimetinib — Cobimetinib will be given orally at 60 mg qd on Days 1-21 of each 28-day treatment cycle

SUMMARY:
In the BRIM-3 trial, which was conducted in patients with previously untreated advanced melanoma harboring the BRAF V600E mutation, vemurafenib, a potent inhibitor of mutated BRAF, was associated with prolonged overall survival (OS) and progression-free survival (PFS) compared to dacarbazine. In the same setting, combined use of vemurafenib and cobimetinib, a selective inhibitor of MEK, yielded a significant improvement in PFS and response rate, compared to vemurafenib monotherapy, along with an advantage in OS, which did not cross the pre-specified significance bounderies (COBRIM trial). In treatment-naïve patients with mutated BRAF, both anti PD-1-based immunotherapy and BRAF-targeted agents are feasible therapeutic options, with the former and latter agents being associated with more durable and earlier responses, respectively.

As suggested by National Comprehensive Cancer Network (NCCN) guidelines, the use of combined BRAF and MEK inhibitors in patients with progressive disease after immunotherapy, is also feasible, but it is not supported by category 1 evidence, in view of the lack of studies conducted in this setting.

The main objective of this phase II trial is to evaluate the efficacy and safety of the combined use of vemurafenib plus cobimetinib in advanced melanoma patients who have received first-line systemic immunotherapy for inoperable locally advanced / metastatic disease.

DETAILED DESCRIPTION:
In the BRIM-3 trial, which was conducted in patients with previously untreated advanced melanoma harboring the BRAF V600E mutation, vemurafenib, a potent inhibitor of mutated BRAF, was associated with prolonged OS and PFS compared to dacarbazine. In the same setting, combined use of vemurafenib and cobimetinib, a selective inhibitor of MEK, yielded a significant improvement in PFS and response rate, compared to vemurafenib monotherapy, along with an advantage in OS, which did not cross the pre-specified significance bounderies (COBRIM trial). In treatment-naïve patients with mutated BRAF, both anti PD-1-based immunotherapy and BRAF-targeted agents are feasible therapeutic options, with the former and latter agents being associated with more durable and earlier responses, respectively.

As suggested by NCCN guidelines, the use of combined BRAF and MEK inhibitors in patients with progressive disease after immunotherapy, is also feasible, but it is not supported by category 1 evidence, in view of the lack of studies conducted in this setting.

The main objective of this phase II trial is to evaluate the efficacy and safety of the combined use of vemurafenib plus cobimetinib in advanced melanoma patients who have received first-line systemic immunotherapy for inoperable locally advanced / metastatic disease.

As evidenced above, vemurafenib inhibits the BRAF V600E kinase, (this mutation is found in 50% to 60% of melanomas), and enables a remarkable clinical response rate, more than 50% and a statistically significant improvement in OS in patients with unresectable stage III and IV melanoma.

However, the clinical utility of BRAF-I treatment is limited by the development of drug resistance. Multiple mechanisms underlie the development of BRAF-I resistance in BRAF V600E melanoma cells including point mutations in MEK1, amplification of mutant BRAF V600E, elevated closely related serinethreonine kinase activity, activating NRAS mutations, increased levels of COT/Tpl2, aberrantly spliced BRAF V600E and growth factor receptor upregulation. Most of these alterations cause BRAF-I resistance by reactivating the MAPK pathway which plays a major role in the proliferation, survival, and metastatic potential of melanoma cells [Shi 2014a, Shi 2014b, Van Allen 2014].

Inhibition of MEK by the novel MEK-I, trametenib or cobimetinib, has been demonstrated to overcome the reactivation of MAPK pathway which is induced by BRAF-I resistance and to increase both OS and OvRR of melanoma patients when combined with BRAF-I [Flaherty 2012a, Flaherty 2012b, Hoeflich 2012, Ribas 2014]. The above-described phase III study, 495 patients with previously untreated unresectable locally advanced or metastatic BRAF V600 mutation-positive melanoma has shown that the combination of vemurafenib and cobimetinib, as compared with vemurafenib alone, resulted in an improvement in PFS and objective responses, with early evidence of improved OS and a somewhat increased toxicity profile [Larkin 2014].

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed, unresectable stage IIIc or stage IV metastatic melanoma, as defined by the American Joint Committee on Cancer 7th edition. Unresectability of stage IIIc disease must have confirmation from a surgical oncologist;
2. Patients with advanced melanoma who have received one prior immunotherapy systemic regimen for advanced disease, for whom vemurafenib/cobimetinib treatment has been scheduled by the treating physician.
3. Adjuvant treatment is allowed, except for anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 agents;
4. Patients must be naïve to treatment for locally advanced unresectable or metastatic with BRAF/MEK inhibitors;
5. Documentation of BRAFV600 mutation-positive status in melanoma tumor tissue BRAF V600 mutation test;
6. At least one measurable lesion according to disease per RECIST v1.1 criteria;
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0- 2;
8. Male or female patient aged ≥ 18 years;
9. Able to participate and willing to give written informed consent prior to performance of any study-related procedures and to comply with the study protocol;
10. Life expectancy ≥ 12 weeks.

Exclusion Criteria:

1. History of any prior systemic treatment for unresectable stage IIIc or stage IV melanoma (prior anti RAF or MEK agents) other than one prior first-line immunotherapy;
2. Palliative radiotherapy within 14 days prior to the first dose of study treatment;
3. Major surgery or traumatic injury within 14 days prior to first dose of study treatment;
4. Patients with active malignancy (other than BRAF- mutated melanoma) or a previous malignancy within the past 3 years are excluded; except for patients with resected melanoma, resected BCC,resected cutaneous SCC, resected melanoma in-situ, resected carcinoma in-situ of the cervix, and resected carcinoma in-situ of the breast; Exclusion Criteria Based on Organ Function.

   Ocular:
5. History of, or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment/central serouschorioretinopathy (CSCR), retinal vein occlusion (RVO) or neovascularmacular degeneration;
6. The risk factors for RVO are listed below. Patients will be excluded if they currently have the following conditions:

   1. Uncontrolled glaucoma with intra-ocular pressures ≥21 mmHg;
   2. Serum cholesterol ≥Grade 2;
   3. Hypertriglyceridemia ≥ Grade 2;
   4. Hyperglycemia (fasting) ≥Grade 2;

   Cardiac:
7. History of clinically significant cardiac dysfunction, including the following:

   1. Current unstable angina;
   2. Symptomatic congestive heart failure of New York Heart Association class 2 or higher;
   3. History of congenital long QT syndrome or mean (average of triplicate measurements) QTcF ≥ 450 msec at baseline or uncorrectable abnormalities inserum electrolytes (sodium, potassium, calcium, magnesium, phosphorus);
   4. Uncontrolled hypertension≥ Grade 2 (patients with a history hypertension controlled with anti-hypertensives to ≤ Grade 1 are eligible);
   5. Left ventricular ejection fraction (LVEF) below institutional lower limit of normal (LLN) or below 50%, whichever is lower.

   Central Nervous System:
8. Patients with active/symptomatic CNS lesions are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Patients enrolled will receive study medication until disease progression, unaccettable toxicity, withdrawal of consent or death, whichever comes first, assested up to 24 month
  OS will be calculated from the first day of treatment until the date of death from any cause.Any patient not know to have died at the time of data analysis will be censored at the time of the last recorded date on which the patient was know to be alive.

SECONDARY OUTCOMES:
PFS | Patients enrolled will receive study medication until disease progression, unaccettable toxicity, withdrawal of consent or death, whichever comes first, assested up to 24 month
  PFS will be defined as the time from initiation of study treatment to the first occurrence of disease progression or death from any cause, whichever occurs first.PFS will be calculated based on disease status evaluated bythe investigator according to RECIST v1.1
ORR | Patients enrolled will receive study medication until disease progression, unaccettable toxicity, withdrawal of consent or death, whichever comes first, assested up to 24 month
  ORR, defined as the proportion of patients with a best overall response of either complete response (CR) or partial response (PR), will be calculated based on disease status evaluated by the investigator accordingto RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Antonio Ascierto, Study Chair — IRCCS Fondazione Pascale Naploli
Locations (1):
- Fondazione G.Pascale, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No